CLINICAL TRIAL: NCT01836796
Title: Metabolic Effects of Dietary Supplementation With Lactobacillus Reuteri DSM 17938 - a Randomised Placebo Controlled Proof-of-concept Study in Type 2 Diabetes
Brief Title: Metabolic Effects of Lactobacillus Reuteri DSM 17938 in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSUB0056
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lactobacillus Reuteri low (Active Comparator): 100 million Lactobacillus Reuteri once daily
  Interventions: Dietary Supplement: Lactobacillus Reuteri; Dietary Supplement: Lactobacillus Reuteri DSM17938
- Lactobacillus Reuteri High (Active Comparator): 10 billion Lactobacillus Reuteri once daily
  Interventions: Dietary Supplement: Lactobacillus Reuteri; Dietary Supplement: Lactobacillus Reuteri DSM17938
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Lactobacillus Reuteri DSM17938

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuteri — 100 million Lactobacillus Reuteri once daily or 10 billion Lactobacillus Reuteri once daily for 12 weeks.
  Arms: Lactobacillus Reuteri High; Lactobacillus Reuteri low
Dietary Supplement: Lactobacillus Reuteri DSM17938 — Powder corresponding to 100 million or 10 billion Lactobacillus Reuteri is added to water once daily for 12 weeks.

SUMMARY:
Recent data suggest that the trillions of bacteria in gastrointestinal tracts (gut microbiota) can function as an environmental factor that modulates the amount of body fat. Obese individuals have an altered gut microbiota and germ-free mice are resistant to developing diet-induced obesity and have lower fasting insulin and glucose concentrations and shows an improved glucose tolerance. Administration of the probiotic bacterium Lactobacillus Gasseri SBT2055 in fermented milk for 12 weeks reduced adiposity and body weight in obese adults possibly by reducing lipid absorption and inflammatory status. However, there are no controlled studies to the investigators knowledge that address whether probiotic supplementation affects glucose metabolism. The investigators hypothesis is that supplementation of Lactobacillus reuteri DSM 17938 may improve metabolic control in type 2 diabetes patients. In addition, the investigators will explore possible mechanisms behind the antihyperglycemic action of Lactobacillus Reuteri.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled randomised study with three parallel groups of type 2 diabetes (T2D) patients receiving either placebo, Lactobacillus reuteri DSM 17938, 1 x 108 (colony-forming units) CFU or Lactobacillus reuteri DSM 17938 CFU 1 x 1010.

The study will be performed at the Clinical Trial Centre (CTC) at the Sahlgrenska University Hospital in Gothenburg. The investigators will recruit forty-five T2D patients of both gender 50-75 yrs, with waist circumference > 80 cm and > 94 cm in women and men, respectively, HbA1c 50-90 mmol/mol and treatment to achieve normoglycemia with lifestyle, insulin with or without oral hypoglycemic agents. Patients who meet all inclusion criteria will be asked to join the study and will be given full written information on the study before being asked to sign a written consent form.

Recruited patients will then undergo a baseline examination with collection of demographic data, fasting blood and urine samples and measurements of blood pressure.

After less than three weeks, the patients return for 1.5 days of investigations. At baseline, urine, blood and faeces samples are taken but also body composition assessed with (Dual Energy X-ray Absorbtion) DEXA, proton magnetic resonance spectroscopy to quantify liver fat content, magnetic resonance imaging (MRI) for determination of visceral adipose tissue and subcutaneous adipose tissue area at the level of L4-L5, a euglycemic hyperinsulinemic clamp at 120 milliunits (mU)/m2/min and finally in conjunction with the glucose clamp, indirect calorimetry, pulse wave analysis and abdominal subcutaneous needle biopsy.

At visit 3 the glucose clamp, day 0, patients will be randomized and given the study medication for the whole study period with instructions to take one dose per day (in the morning before breakfast). Patients then return at day 28 and day 56 for urine, faeces and blood sampling. After 12 weeks supplementation on day 84±7 days, blood, urine and faeces samples and all procedures performed at baseline in conjunction with day 0 are repeated. Moreover, patients return study medications not being used. Finally, patients who completed the study and will be asked to book a visit to their ordinary diabetes team.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with a duration > 6 months
* Adults 50- 75 years of age
* Abdominal obesity (females waist > 80 cm; males waist > 94 cm)
* HbA1c 50-90 mmol/mol
* Anti-hyperglycemic treatment with lifestyle, oral agents and insulin
* Written informed consent
* Stated availability throughout the study period
* Fasting C-peptide > 0.27 nmol/l
* BMI 25-40 kg/m2
* Stable weight (± 5 kg) and HbA1c (± 5 mmol/mol) for 6 months

Exclusion Criteria:

* Autoimmune diabetes eg type 1 diabetes
* Psychiatric illness e g claustrophobia or alcoholism, cancer diagnosis and no foreseeable need of treatment with corticosteroids or antibiotics under the 12 week study period
* Heavy nicotine users suggesting abstinence problems during the clamp
* Anti-coagulation with warfarin
* Ischemic heart disease with an event < 6 months ago
* Inflammatory bowel disease
* Administration of antibiotics 4 weeks before inclusion
* Administration of probiotics 2 weeks before inclusion
* Participation in other clinical trials
* Other medical conditions, as judged by the screening doctor, that might jeopardize compliance to the protocol eg severe obesity interfering with access to peripheral veins
* Pregnancy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks compared to baseline

SECONDARY OUTCOMES:
Liver steatosis | Baseline compared to 12 weeks
Insulin sensitivity in muscle, liver and adipose tissue | Baseline compared to 12 weeks
Urine albumine excretion rate | Baseline compared to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Centre, Gröna Stråket 12, Sahlgrenska University Hospital, Gothenburg, Sweden